CLINICAL TRIAL: NCT00896883
Title: A Prospective, Non-Randomized, Limited-Use Evaluation of the Middle Turbinate Implant for Affixing the Middle Turbinate to the Nasal Septum
Brief Title: Evaluation of the Middle Turbinate Implant for Affixing the Middle Turbinate to the Nasal Septum
Acronym: MTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ENTrigue Surgical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CSA2008-02
Record Dates: First submitted 2009-05-08; First posted 2009-05-12 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Sinusitis
Keywords: turbinate; implant; sinus surgery; Turbinates
MeSH Terms: conditions — Sinusitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Middle Turbinate Implant (Experimental): Subjects to receive Middle Turbinate Implant
  Interventions: Device: Middle Turbinate Implant

INTERVENTIONS:
Device: Middle Turbinate Implant — Middle Turbinate Implant placement at time of surgery and follow ups.
  Other Names: MTI

SUMMARY:
The purpose of this study is to determine the functional performance of the Middle Turbinate Implant (MTI). The MTI will be used in all patients requiring endoscopic sinus surgery in which the Principal Investigator determines clinical relevance.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between the ages of 18 and 65 years and will be receiving endoscopic sinus surgery.
* Subject is able to provide a signed informed consent form.
* Subject will agree to comply with all study-related procedures.
* Subject is not pregnant at this time by confirmation of one of the following:

  * Subject is male
  * Subject not of child bearing age
  * Subject is surgically sterile
  * Subject is not pregnant per negative hCG test
  * Subject does not plan on becoming pregnant and is not breast feeding during the course of the study.

Exclusion Criteria:

* Subject does not meet inclusion criteria.
* Presence of non-viable tissue at the implantation site.
* History of septal perforation.
* History of polyps.
* Presence of concha bullosa.
* Subject is currently using CPAP (Continuous Positive Airway Pressure) for sleep apnea.
* Subject is participating in a clinical trial which could affect the healing of the middle turbinate.
* Subject has uncontrolled diabetes.
* Subject is a:

  * smoker
  * severe drug abuser
  * severe alcohol abuser
* Subject has an autoimmune disease deemed clinically significant by the Principal Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-04; Primary Completion 2009-11 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Functional performance of the MTI | 1 month

SECONDARY OUTCOMES:
Visual tissue reaction to the Middle Turbinate Implant | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Ronald B Kuppersmith, MD, Principal Investigator — Texas ENT and Allergy
Locations (4):
- United States (4):
  - Becker Nose and Sinus Center, Sewell, New Jersey
  - Texas Sinus Center, Boerne, Texas
  - Texas ENT and Allergy, College Station, Texas
  - San Antonio Ear, Nose and Throat Research, San Antonio, Texas